CLINICAL TRIAL: NCT02430350
Title: Compound Edaravone Injection for Acute Ischemic Stroke, a Multi-center, Randomized, Double-blind, Parallel, and Active-controlled PhaseⅢTrial
Brief Title: Study of Compound Edaravone Injection for Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-23-02
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compound Edaravone (Experimental): Compound Edaravone Injection 37.5mg/dose (Edaravone 30mg, (+)-Borneol 7.5mg), one dose every 12 hours, continue for 14 days
  Interventions: Drug: Compound Edaravone Injection
- Edaravone (Active Comparator): Edaravone Injection 30 mg/dose, one dose every 12 hours, continues for 14 days
  Interventions: Drug: Edaravone Injection

INTERVENTIONS:
Drug: Compound Edaravone Injection
  Arms: Compound Edaravone
Drug: Edaravone Injection
  Arms: Edaravone

SUMMARY:
The primary objective of the study is to confirm the efficacy of compound Edaravone Injection via intravenous infusion every 12 hours in the patients with Acute Ischemic Stroke(AIS) in a double-blind, active-controlled manner. The study is also to examine the safety of compound Edaravone Injection for the AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients, diagnosed of ischemic stroke;
* Onset of stroke is less than or equal to 48 hours;
* There are clear signs of neurological deficit: 4≤NIHSS score≤24, and also, the sum of NIHSS score for the upper limb and the lower limb is greater than or equal to 2;
* Patients signed written inform consent

Exclusion Criteria:

* Cranial CT scan finds intracranial bleeding disorders: hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage;
* Iatrogenic stroke;
* Severe disturbance of consciousness: NIHSS category 1a for consciousness is greater than 1；
* The mRS score prior to this onset is greater than 1;
* Transient ischemic attack (TIA);
* SBP after blood pressure control is still greater than or equal to 220 mmHg, or DBP after blood pressure control is still greater than or equal to 120 mmHg;
* Patients with severe mental disorders and dementia;
* ALT or AST is greater than 2.0×ULN or previously known liver diseases, such as acute hepatitis, chronic active hepatitis, liver cirrhosis;
* Serum Creatinine (SCr) is greater than 1.5×ULN, Creatinine Clearance (CrCl) is less than 50 ml/min or previously known severe renal diseases;
* Therapeutic neuroprotective agents have been applied after onset of stroke, including commercially available edaravone, nimodipine, ganglioside, citicoline, piracetam, butyl benzene peptides, Urinary Kallidinogenase;
* Arterial or venous thrombolytic therapy has been applied after onset of stroke;
* Patients with malignant tumors or receiving concurrent antitumor treatment;
* Patients with severe systemic disease, life expectancy is less than 90 days;
* allergic to edaravone , (+)-Borneol or related excipients;
* Pregnant or lactating women;
* Have major surgery within 4 weeks before enrollment;
* Participated in other clinical studies within 30 days before randomization; or participating in other clinical trials at present;
* The investigators consider the patients are not suitable for this trial.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with mRS ≤1 on day 90 | day 90

SECONDARY OUTCOMES:
mRS score on day 90 | day 90
Changes of NIHSS score from baseline on day 14 | day 14
The proportion of patients with NIHSS score 0-1 (including motor function) on day 14, 30, 90 | day 14, 30, 90
The proportion of patients with Barthel Index (BI) score greater than or equal to 95 on day 14, 30, 90 | day 14, 30, 90
Montreal Cognitive Assessment(MoCA) score on day 14, 30, 90 | day 14, 30, 90
Stroke Impact Scale (SIS) score on day 90 | day 90

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (48):
- China (48):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Navy General Hospital of The Chinese PLA, Beijing, Beijing Municipality
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Nanning Second People's Hospital, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Second Affiliated Hospital of Haerbin Medical University, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The Third Affiliated Hospital of Inner Mongolia Medical University, Baotou, Inner Mongolia
  - Central Hospital of Baotou, Baotou, Inner Mongolia
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Huai'an First Affiliated Hospital of Nanjing Medical University, Huai'an, Jiangsu
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongda Hospital,Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Yangzhou No.1 People's Hospital, Yangzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The Forth Hospital of Jilin University, Siping, Jilin
  - Siping Central Hospital, Siping, Jilin
  - The General Hospital of Shenyang Military, Chinese PLA, Shenyang, Liaoning
  - The Sceond Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Yangpu Hospital, Tongji University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Lishui People's Hospital, Lishui, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu J, Wang A, Meng X, Yalkun G, Xu A, Gao Z, Chen H, Ji Y, Xu J, Geng D, Zhu R, Liu B, Dong A, Mu H, Lu Z, Li S, Zheng H, Chen X, Wang Y, Zhao X, Wang Y; TASTE Trial Investigatorsdagger. Edaravone Dexborneol Versus Edaravone Alone for the Treatment of Acute Ischemic Stroke: A Phase III, Randomized, Double-Blind, Comparative Trial. Stroke. 2021 Mar;52(3):772-780. doi: 10.1161/STROKEAHA.120.031197. Epub 2021 Feb 16. PMID 33588596